CLINICAL TRIAL: NCT06135714
Title: a Randomized Trial for OLIGo Metastases Breast cAncer With or Without Metastasis-dIrected Therapy
Brief Title: Metastasis-directed Therapy for Oligometastases of Breast Cancer
Acronym: OLIGAMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Principal Investigator, Toshiyuki Ishiba, M.D.Ph.D., Assistant professor, Tokyo Medical and Dental University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG2110
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Oligometastasis; Metastatic Breast Cancer
Keywords: SBRT; Surgery; Stereotactic Body Radiation Therapy; Metastasis-directed Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: If this 12-week systemic therapy does not cause any progression or complete response, patients proceed to second registration for randomization; arm A continues same systemic therapy alone, and arm B performs MDT followed by same systemic therapy. The MDT will involve either RT or surgery, and RT will involve mainly SBRT and partly conventional RT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Standard of care (Placebo Comparator): Continuation of systemic drug therapy.
  Interventions: Drug: Systemic therapy for 12 weeks after primary registration; Drug: Same systemic therapy after secondary registration
- Arm B: Metastasis-directed therapy followed by Standard of care (Experimental): Metastasis-directed therapy (radiation or surgery for oligometastasis) + systemic drug therapy.
  Interventions: Drug: Systemic therapy for 12 weeks after primary registration; Procedure: Radiation therapy (SBRT/conventional RT); Procedure: Surgery; Drug: Same systemic therapy after secondary registration

INTERVENTIONS:
Drug: Systemic therapy for 12 weeks after primary registration — * Luminal BC
    1. Denovo stage IV
       Premenopausal(PRE): Aromatase inhibitor(AI) + CDK4/6 inhibitor(CDK) +LHRH agonist, or Fulvestrant(FUL) + CDK4/6 inhibitor +LHRH agonist
       Postmenopausal(POST): AI + CDK
    2. Recurrence after completion of postoperative endocrine therapy
       PRE: AI + CDK +LHRH agonist, or FUL + CDK +LHRH agonist
       POST: AI + CDK, or FUL + CDK
    3. Recurrence during postoperative endocrine therapy
       PRE: FUL + CDK +LHRH agonist, or AI + CDK +LHRH agonist
       POST: FUL + CDK
  * HER2-positive BC
  Pertuzumab + Trastuzumab + Taxane (docetaxel or paclitaxel)
  ・Triple negative BC.
  1. PD-L1 negative - following a) or b)
     1. Taxane (naive for taxane)
     2. S-1 or Capecitabine or Eriblin (previously treated with taxane)
  2. PD-L1 positive - following a) or b)
     1. Pembrolizumab + Gemcitabine + Carboplatin
     2. Atezolizumab + Nab-paclitaxel
  3. BRCA-mutation positive Olaparib
Procedure: Radiation therapy (SBRT/conventional RT) — Brain: 18-24Gy/1Fr. or 27Gy/3Fr. or 30Gy/5Fr. Lung: 42Gy/4Fr.(peripheral) or 50Gy/8Fr.(central) or 60Gy/25Fr.(ultra central) Liver/Adrenal: 40Gy/5Fr. Bone: 35Gy/5Fr. Distant lymph node: 45/10Fr. or 60Gy/25Fr.
  Arms: Arm B: Metastasis-directed therapy followed by Standard of care
Procedure: Surgery — Surgery for the oligometastases
  Arms: Arm B: Metastasis-directed therapy followed by Standard of care
Drug: Same systemic therapy after secondary registration — * Luminal BC
    1. Denovo stage IV
       Premenopausal(PRE): Aromatase inhibitor(AI) + CDK4/6 inhibitor(CDK) +LHRH agonist, or Fulvestrant(FUL) + CDK4/6 inhibitor +LHRH agonist
       Postmenopausal(POST): AI + CDK
    2. Recurrence after completion of postoperative endocrine therapy
       PRE: AI + CDK +LHRH agonist, or FUL + CDK +LHRH agonist
       POST: AI + CDK, or FUL + CDK
    3. Recurrence during postoperative endocrine therapy
       PRE: FUL + CDK +LHRH agonist, or AI + CDK +LHRH agonist
       POST: FUL + CDK
  * HER2-positive BC
  Pertuzumab + Trastuzumab + Taxane (docetaxel or paclitaxel)
  ・Triple negative BC.
  1. PD-L1 negative - following a) or b)
     1. Taxane (naive for taxane)
     2. S-1 or Capecitabine or Eriblin (previously treated with taxane)
  2. PD-L1 positive - following a) or b)
     1. Pembrolizumab + Gemcitabine + Carboplatin
     2. Atezolizumab + Nab-paclitaxel
  3. BRCA-mutation positive Olaparib

SUMMARY:
OLIGAMI trial is a multi-institutional, two-arm, open-label, randomized controlled phase III trial being conducted with the participation of 50 hospitals belonging to Japan Clinical Oncology Group. After the first registration, all patients will be performed in a 12-week, subtype-specific, systemic therapy consisting of CDK4/6 inhibitors with hormonal therapy for luminal BC, docetaxel with trastuzumab and pertuzumab for HER2-positive BC, chemotherapy with immune checkpoint inhibitors for triple-negativeBC expressing PD-L1, and olaparib for cases harboring BRCA mutations. For other triple-negative BC, chemotherapy will be administered. If this 12-week systemic therapy does not cause any progression or complete response, patients proceed to second registration for randomization; arm A continues same systemic therapy alone, and arm B performs MDT followed by same systemic therapy. The MDT will involve either RT or surgery, and RT will involve mainly SBRT and partly conventional RT.

DETAILED DESCRIPTION:
A brief background discussion: Oligometastases were initially described as a concept bridging localized disease with widespread distant metastases, but a consensus on its definition has yet to be reached. Recently, the term "metastasis-directed therapy" (MDT) was coined to encompass local therapy for distant metastases, including surgery and radiation therapy (RT), especially stereotactic body radiation therapy (SBRT). Though OLIGO-BC1 and SABR-COMET have indicated the potential benefits of MDT for oligometastases , NRG-BR002 revealed no significant difference in progression-free survival (PFS). As a definitive conclusion to this clinical question has not been reached, there is an increasing demand for phase III trials focusing on breast cancer (BC). We planned the JCOG2110, also called as OLIGAMI trial. Trial design: OLIGAMI trial is a multi-institutional, two-arm, open-label, randomized controlled phase III trial being conducted with the participation of 50 hospitals belonging to Japan Clinical Oncology Group. After the first registration, all patients will be performed in a 12-week, subtype-specific, systemic therapy consisting of CDK4/6 inhibitors with hormonal therapy for luminal BC, docetaxel with trastuzumab and pertuzumab for HER2-positive BC, chemotherapy with immune checkpoint inhibitors for triple-negativeBC expressing PD-L1, and olaparib for cases harboring BRCA mutations. For other triple-negative BC, chemotherapy will be administered. If this 12-week systemic therapy does not cause any progression or complete response, patients proceed to second registration for randomization; arm A continues same systemic therapy alone, and arm B performs MDT followed by same systemic therapy. The MDT will involve either RT or surgery, and RT will involve mainly SBRT and partly conventional RT. Eligibility criteria: OLIGAMI trial will encompass all subtypes of advanced BC. The key criteria of the first registration are as follows: 1) Histologically diagnosed as invasive BC. Biopsy from oligometastases is desirable but not required. 2) Diagnosed with advanced BC with oligometastases by neck to pelvis enhanced CT, FDG-PET,and brain enhanced MRI. 3) Oligometastases defined as: (i) Maximum diameter of each tumor is 3 cm or less. (ii) Total number of 3 or less. (iii) In case of brain metastasis, maximum diameter is 2 cm or less and asymptomatic. 4) The patient with local recurrence is included. 5) De novo stage IV BC is included. The criteria of secondary registration are as follows: 1) The planned number of courses of systemic therapy has been performed. 2) No progression or new distant metastasis by response evaluation. 3) At least one oligometastasis remains. Specific Aims: OLIGAMI trial aims to confirm the superiority of MDT to systemic therapy for oligometastases of BC. The primary endpoint is overall survival (OS) after randomization, while the secondary endpoints include OS after first registration, PFS, progression site (oligometastases vs. non-oligometastases), PFS specifically related to MDT (restricted arm B), proportion of adverse events and serious adverse events, and the non-progression proportion of health-related quality of life. Statistical methods: The sample size was calculated as 268 to detect 12% of 5-year OS difference with a one-sided alpha of 0.05, power of 70%, 3 years of accrual, and 5 years of follow up. Therefore, we assumed the planned sample size for second registration for randomization as 270. We set the number of first registration as 340, assuming that there may be some patients with progression or complete response after the systemic therapy for 12 weeks. Present accrual and target accrual: The patient accrual will start in November 2023. Enrolment of 340 patients for first registration is planned over a 3-year accrual period.

ELIGIBILITY:
Primary Registration Eligibility Criteria:

1. Histologically diagnosed as invasive breast cancer. Biopsy from oligometastasis is desirable but not required.
2. Histologically proven positive/negative for ER, PgR, and HER2, and classified as luminal, HER2-positive, or TN breast cancer.
3. One of the following <1> to <4>; <1>In case of no history of breast cancer in the past, either (i) or (ii) below.

   (i) Unilateral noninvasive breast cancer at registration, diagnosed as invasive breast cancer by biopsy from oligometastasis (ii) Unilateral invasive breast cancer at registration <2>In case of having a history of mastectomy or breast-conserving surgery for unilateral noninvasive breast cancer, either (i) or (ii) below. (i) Absence of breast/chest wall tumor at registration and diagnosed as invasive breast cancer by biopsy from oligometastasis (ii) Unilateral invasive breast cancer at registration (whether ipsilateral or contralateral to previous breast cancer) <3>In case of having a history of mastectomy or breast-conserving surgery for unilateral invasive breast cancer, either (i) or (ii) below. (i) Absence of breast/chest wall tumor at registration (ii) Ipsilateral invasive/noninvasive breast cancer to previous breast cancer at registration and diagnosed as recurrence <4>In case of having a history of mastectomy or breast-conserving surgery for unilateral noninvasive breast cancer and contralateral invasive breast cancer, no breast/chest wall tumor at registration.
4. Diagnosed with advanced breast cancer with oligometastasis by neck to pelvis enhanced CT, FDG-PET (PET/CT), and brain enhanced MRI.
5. oligometastasis defined as: (i) Maximum diameter of each tumor is 3 cm or less (ii) Total number of 3 or less. (iii) In case of brain metastasis, maximum diameter is 2 cm or less and asymptomatic.
6. No distant metastasis other than oligometastasis.
7. Metastasis-directed therapy (radiation or surgery) is considered feasible for all oligometastases.
8. In case of bone metastasis, none of the following:

   (i) Metastasis of three consecutive vertebral bodies (ii) Spinal metastasis extending into the spinal canal (Bilsky grade is 1b or higher) (iii) Long bone metastasis extending to the femoral head, neck, and trochanter (iv) Long bone metastasis with more than 1/3 of bone cortical defects (v) Severe pain uncontrolled with drugs.
9. Aged 18-80 years.
10. ECOG performance status of 0 or 1.
11. A measurable lesion is not required.
12. No history of surgery, drug therapy, or radiotherapy for distant metastasis. Bisphosphonate preparations and RANKL inhibitors before registration, and surgery for the purpose of diagnosing metastasis are permitted.
13. No radical surgery of the primary tumor or regional lymph nodes between diagnosis of oligometastasis to registration.
14. In the case of recurrent breast cancer, disease-free interval of 12 months or more from surgery, perioperative chemotherapy, or molecular targeted therapy for initial treatment of breast cancer.
15. No prior treatment of endocrine therapy, chemotherapy, molecular targeted therapy, and immunotherapy against any other malignancies within 5 years.
16. Adequate organ function within 14 days prior to the first registration. (i) ANC >= 1500 cells/mm3 (ii) Hemoglobin >= 9.0 g/dL (iii) Platelet count >= 100,000/ mm3 (iv) Serum bilirubin <= 1.5 mg/dL (v) AST <= 100 U/L (vi) ALT <= 100 U/L (vii) Creatinine <= 1.5 mg/dL (<= 2.3 mg/dL for luminal breast cancer)
17. Ejection fraction of cardiac function is defined over 50%.
18. Written informed consent.

Secondary Registration Eligibility Criteria:

1. Primary registration in this study, and the planned number of courses of systemic drug therapy by subtype has been performed.
2. No progression or new distant metastasis by response evaluation.
3. Secondary registration is within 28 days from response evaluation.
4. Within 84-126 days from the primary registration.
5. At least one oligometastasis remains on imaging and considered feasible to definitive local therapy.
6. No metastasis-directed therapy for breast cancer after primary registration.
7. ECOG performance status of 0 or 1.
8. Adequate organ function within 14 days prior to the second registration. (i) ANC >= 1500 cells/mm3 (ii) Hemoglobin >= 9.0 g/dL (iii) Platelet count >= 100,000/ mm3 (iv) Serum bilirubin <= 1.5 mg/dL (v) AST <= 100 U/L (vi) ALT <= 100 U/L (vii) Creatinine <= 1.5 mg/dL (<= 2.3 mg/dL for luminal breast cancer)

Exclusion Criteria:

1. Active malignancies curatively treated with no evidence of disease for >= 5 years prior to randomization.
2. Infection with care.
3. Fever up 38 degrees Celsius.
4. Childbearing potential, delivery after 28 days, breastfeeding
5. Mental disorders.
6. Continuously take steroids or immunosuppressive drugs.
7. Unstable angina or history of cardiac infarction within 6months.
8. Uncontrolled Hypertension.
9. Uncontrolled Diabetes mellitus.
10. Congestive heart failure deserved class II of New York Heart Association (NYHA), uncontrolled Dilated or Hypertrophic cardiomyopathy.
11. Severe arrhythmia need to cure (except Atrial fibrillation, Paroxysmal supraventricular tachycardia)
12. Interstitial pneumonia, pulmonary fibrosis, severe emphysema diagnosed chest CT scan.
13. HBs Ag+

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival after second registration | 5 years

SECONDARY OUTCOMES:
Overall survival after primary registration | 5 years
Progression-free survival | 5 years
Progression site (oligometastasis, lesion other than oligometastasis) | 5 years
Oligometastatic progression-free survival for each definitive local therapy (group B only) | 5 years
Adverse event rate | 5 years
Serious adverse event rate | 5 years
HR-QOL non-worsening rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Toshiyuki Ishiba, M.D.Ph.D., Principal Investigator — Tokyo Medical and Dental University; Tadahiko Shien, M.D.Ph.D., Study Chair — Okayama University; Ikuno Nishibuchi, M.D.Ph.D., Principal Investigator — Hiroshima University; Fumitaka Hara, M.D.Ph.D., Principal Investigator — The Cancer Institute Hospital of Japanese Foundation for Cancer Research; Naoto Shikama, M.D.Ph.D., Study Chair — Juntendo University
Locations (1):
- Tokyo Medical and Dental Univetsity, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Background] Sasaki K, Ishiba T, Nishibuchi I, Hara F, Sekino Y, Machida R, Shibata T, Kawahara D, Sagara Y, Naito Y, Terata K, Ozaki Y, Shimomura A, Sakai T, Shigematsu H, Sudo K, Nozawa K, Yoshimura M, Shikama N, Mizowaki T, Shien T. A randomized controlled trial of metastasis-directed therapy for oligometastases in breast cancer: OLIGAMI trial (JCOG2110). Jpn J Clin Oncol. 2026 Jan 30:hyag019. doi: 10.1093/jjco/hyag019. Online ahead of print. PMID 41615067
- See also: Related Info — https://jcog-breast.com/report/now/jcog2110/